CLINICAL TRIAL: NCT04973254
Title: Cabotegravir-Rilpivirine Long Acting (CAB-RPV LA) Implementation Strategies Among High-Risk Populations
Brief Title: Improving Treatment and Retention Adherence in Nontraditional Settings
Acronym: I-TRAINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-41724; 4300844001 (Other Grant/Funding Number: ViiV Healthcare)
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections
Keywords: HIV injectable medication; Cabotegravir-Rilpivirine Long Acting (CAB-RPV LA); Treatment adherence; Community-based delivery strategy; Patient-centeredness; Acceptability; Feasibility
MeSH Terms: conditions — HIV Infections; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Three-arm cohort study comparing adherence to HIV treatment of monthly injections delivered outside of standard clinical settings to treatment adherence in the HIV clinic setting and to HIV standard care delivered in the HIV clinic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1- HIV injection at a community-based site (Experimental): CAB-RPV LA administered to patients in an alternative community-based site
  Interventions: Other: CAB-RPV LA
- Cohort 2- HIV injection at a HIV clinic (Active Comparator): CAB-RPV LA administered to patients in the HIV clinic
  Interventions: Other: CAB-RPV LA
- Cohort 3- Standard of care for HIV (Active Comparator): Individuals who share characteristics of cohort 1 and are engaged in standard of care
  Interventions: Other: Standard treatment within an HIV clinic

INTERVENTIONS:
Other: CAB-RPV LA — Monthly administration of injectable HIV medication
  Other Names: Cabotegravir-Rilpivirine Long Acting
  Arms: Cohort 1- HIV injection at a community-based site; Cohort 2- HIV injection at a HIV clinic
Other: Standard treatment within an HIV clinic — Standard of care for HIV positive patients will be provided in the HIV clinic that may include HIV medication or may include oral medications.
  Arms: Cohort 3- Standard of care for HIV

SUMMARY:
This is a hybrid implementation-effectiveness study using both qualitative and quantitative methods. The research aims to examine whether providing a new, but approved, HIV once a month injection treatment [Cabotegravir-Rilpivirine Long Acting (CAB-RPV LA)] to individuals who are living with HIV outside of the standard doctors office or clinic increases adherence to treatment. This HIV monthly injections treatment which is already being delivered within the clinic setting, will be administered to participants in community partner spaces, reducing the barriers that having to present to a traditional clinic for treatment creates.

Individuals who will receive the injection need to have a history of being unable to take their HIV oral medication, as well as other barriers to care that make it difficult to engage in a traditional clinic setting. These barriers may include, but are not limited to, homelessness, substance use, mental illness, and stigma around their diagnosis.

Data will be collected on whether it was easier for the participants to receive care in a non-traditional setting, as well as whether the injection made it easier for them to remain adherent to their HIV medication in comparison to standard oral HIV medication.

DETAILED DESCRIPTION:
The proposed implementation research is designed to evaluate a novel approach to engage individuals with HIV who are at the highest risk for not accessing care or adhering to treatment. The investigators are not testing CAB-RPV LA; this is an approved drug. The investigators are also not studying the drug nor studying it for a new population, new dosage or new route of administration. Rather, the investigators are conducting an implementation three-arm cohort study that uses quantitative methods and propose to test implementation of CAB-RPV LA in community-based settings. The three cohorts/groups will be:

* cohort 1- individuals who receive CAB-RPV LA at an alternative community-based site
* cohort 2- individuals who receive CAB-RPV LA in the HIV clinic
* cohort 3- individuals who share characteristics of cohort 1 and are engaged in standard of care

The research is designed to answer the following implementation and clinical questions.

A. Implementation Questions

1. Will community-based delivery of CAB-RPV LA be an acceptable and feasible delivery method to high-risk people living with HIV (PLWH) from the patient, provider and community organization perspectives? (acceptability/feasibility)
2. Can a community-based delivery strategy lead to initiation and completion of injections for six months for at least 80% of individuals who are enrolled into cohort 1 for an initial visit in an outreach setting? (reach) See Section 11 for information on the details of the sample size calculations and Section 7.2 for how study staff will stay in contact with participants to maximize potential for longer term engagement.
3. What are the characteristics of patients who are most likely to have an initial injection and do these characteristics differ for individuals who receive CAB-RPV LA in and outside of the HIV clinic? (equity)
4. Are patients who are seen for CAB-RPV LA in community-based settings satisfied with their HIV care? (patient-centeredness)
5. Will consistent delivery of CAB-RPV LA be possible in community-based (non-HIV clinic) settings? (feasibility)
6. Will the providers at a drop-in center or community-based organization be willing to implement CAB-RPV LA within their non-traditional setting? (adoption)

B. Clinical Questions

1. Can individuals targeted for intervention at community-based delivery site achieve viral suppression and receive initial injection?
2. Can a community-based delivery strategy ensure engagement in services and receipt of CAB-RPV LA visits among high-risk populations? (effectiveness)
3. Is a community-based delivery strategy using CAB-RPV LA superior to the current standard of care in ensuring treatment adherence for individuals at highest risk? (effectiveness) Can high-risk individuals who receive community-based CAB-RPV LA be adherent to care, defined as undetectable viral load, for six months?

ELIGIBILITY:
Inclusion Criteria for Cohort 1:

* HIV-positive
* English or Spanish speaking
* Lab values that indicate the patient is a candidate for the medication and virally suppressed
* Willing to complete the locator form to receive appointment reminders prior to follow-up data collection

Inclusion Criteria for Cohort 2:

* HIV-positive
* English or Spanish speaking
* Enrolled in care and receiving CAB-RPV LA injection at Boston Medical Center Infectious Disease Clinic (HIV clinic)
* Willing to complete the locator form to receive appointment reminders prior to follow-up data collection

Inclusion Criteria for Cohort 3:

* HIV-positive
* English or Spanish speaking
* Enrolled in care but NOT receiving CAB-RPV LA injection at Boston Medical Center Infectious Disease Clinic (HIV clinic)
* Willing to complete the locator form to receive appointment reminders prior to follow-up data collection
* Matched to participants demographically and in terms of other characteristics in Cohort 1 at a 2:1 ratio

Exclusion Criteria (for all 3 cohorts unless stated):

* Not virally suppressed prior to beginning CAB-RPV LA (does not apply to cohort 3)
* A history of adhering fully to their antiretroviral therapy (ART)
* Not willing to take CAB-RPV LA after detailed discussion of what the use of CAB-RPV LA will entail (does not apply to cohort 3)
* Unable to undergo clinical eligibility testing to confirm eligibility (does not apply to cohort 3)
* A history of integrase inhibitor mutations suggesting resistance to Cabotegravir or Cabenuva
* A history or evidence of resistance to either integrase strand transfer inhibitor (INSTI) or non-nucleoside reverse transcriptase inhibitors (NNRTI) HIV drugs
* Currently pregnant or breastfeeding
* Currently has HIV 1 with an HIV 2 co-infection or an HIV 2 infection
* Taking any drugs that have known interactions with Cabenuva, including but not limited to carbamazepine, oxcarbazepine, phenobarbital, phenytoin, St Johns Wort, systemic Dexamethasone, rifabutin, rifampin and rifapentine
* Chronic Hepatitis B infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mari-Lynn Drainoni, PhD, Principal Investigator — BU School of Medicine, Infectious Diseases and Boston Medical Center
Locations (2):
- United States (2):
  - Boston Medical Center, Center for Infectious Disease, Boston, Massachusetts
  - Boston Medical Center, Project Trust, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1- HIV Injection at a Community-based Site | Cohort 2- HIV Injection at a HIV Clinic | Cohort 3- Standard of Care for HIV
Started | 5 | 18 | 2
Completed | 5 | 17 | 2
Not Completed | 0 | 1 | 0
Not completed — Not adherent | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1- HIV Injection at a Community-based Site | Cohort 2- HIV Injection at a HIV Clinic | Cohort 3- Standard of Care for HIV | Total
Number analyzed (Participants) | 5 | 18 | 2 | 25
Age, Continuous [Median (Full Range); unit: years] | 36 [33 to 45] | 45 [39 to 62] | 53.5 [47 to 60] | 46 [33 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 0 | 8
  Male | 4 | 11 | 2 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 8 | 0 | 8
  Asian | 0 | 2 | 0 | 2
  Hispanic or Latino | 0 | 6 | 1 | 7
  White | 4 | 0 | 1 | 5
  Other | 1 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 18 | 2 | 25

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Cabenuva Injections
Description: The number of participants who received CAB-RPV LA injections within the treatment window.
Time Frame: 3 months, 6 months
Population: Data were only analyzed for Cohorts 1 and 2 for this outcome measure since the 2 participants in Cohort 3 never came in for a study visit so no data were collected.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3- Standard of Care for HIV: Individuals who share characteristics of cohort 1 and are engaged in standard of care.
  Standard of care for HIV positive patients will be provided in the HIV clinic that may include HIV medication or may include oral medications.
Arm/Group | Cohort 1- HIV Injection at a Community-based Site | Cohort 2- HIV Injection at a HIV Clinic | Cohort 3- Standard of Care for HIV
Number analyzed (Participants) | 5 | 18 | 0
Participants
  3 months | 1 | 17 | 0
  6 months | 1 | 17 | 0

2. Primary Outcome: Adherence to Primary Care Appointments
Description: The number participants who had a primary care appointment in the previous 3 months.
Time Frame: 3 months, 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- HIV Injection at a Community-based Site | Cohort 2- HIV Injection at a HIV Clinic | Cohort 3- Standard of Care for HIV
Number analyzed (Participants) | 5 | 17 | 0
Participants
  3 months | 5 | 17 | 0
  6 months | 2 | 16 | 0

3. Primary Outcome: Adherence to Mental Health/Behavioral Appointments
Description: The number participants who had a mental health/behavioral appointment in the previous 3 months.
Time Frame: 3 months, 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3- Standard of Care for HIV: Individuals who share characteristics of cohort 1 and are engaged in standard of care, Standard of care for HIV positive patients will be provided in the HIV clinic that may include HIV medication or may include oral medications.
Arm/Group | Cohort 1- HIV Injection at a Community-based Site | Cohort 2- HIV Injection at a HIV Clinic | Cohort 3- Standard of Care for HIV
Number analyzed (Participants) | 5 | 17 | 0
Participants
  3 months | 2 | 4 | 0
  6 months | 1 | 3 | 0

4. Primary Outcome: Adherence to Substance Abuse Appointments in Cohorts 1 and 2
Description: The number participants who had a substance abuse appointment in the previous 3 months.
Time Frame: 3 months, 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1- HIV Injection at a Community-based Site | Cohort 2- HIV Injection at a HIV Clinic | Cohort 3- Standard of Care for HIV
Number analyzed (Participants) | 5 | 17 | 0
Participants
  3 months | 5 | 0 | 0
  6 months | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cohort 1- HIV Injection at a Community-based Site | Cohort 2- HIV Injection at a HIV Clinic | Cohort 3- Standard of Care for HIV
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/17 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/17 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/17 | 0/2

LIMITATIONS AND CAVEATS:
There were challenges enrolling participants resulting in only 25 actual participants from the anticipated enrollment of 100, with only 2 participants in Cohort 3. However, after the 2 participants in Cohort 3 were enrolled they did not participate in the study and no data were collected on them which is why there are no results for Cohort 3. Results for the outcome measures are provided for Cohort 1 (n=5) and Cohort 2 (n=18).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT04973254/Prot_SAP_000.pdf